CLINICAL TRIAL: NCT06859203
Title: Prospective Evaluation of Fluciclovine (18F) PET/CT in Patients with Prior Negative PSMA PET/CT
Brief Title: A Prospective, Bicentric Evaluation of Fluciclovine PET-imaging in Patients with Prior Negative or Inconclusive PSMA-ligand PET
Acronym: REFINE
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-643-S-NP
Record Dates: First submitted 2025-02-27; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Biochemical Recurrence of Malignant Neoplasm of Prostate
Keywords: prostate cancer; biochemical recurrence; PET; PSMA; fluciclovine; BCR; prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- Prostate cancer patients with biochemical recurrence after negative/inconclusive PSMA PET/CT: This cohort comprises male patients with biochemically recurrent prostate cancer following definitive treatment-such as surgery or radiotherapy-who have previously undergone a PSMA PET/CT scan that was either negative or inconclusive. The primary intervention of interest is the fluciclovine (18F) PET/CT scan, which is performed as part of their routine clinical care to detect sites of recurrent disease.

SUMMARY:
The REFINE study is evaluating whether a fluciclovine (18F) PET/CT scan can detect recurrent prostate cancer in patients whose previous PSMA PET/CT was negative or inconclusive.

DETAILED DESCRIPTION:
The REFINE study is a prospective, bicentric observational trial conducted at two specialized nuclear medicine centers in Germany to evaluate the technical performance of fluciclovine (18F) PET/CT imaging in a real-world clinical setting. Patients with prostate cancer recurrence after definitive treatment who previously underwent a negative or inconclusive PSMA PET/CT are enrolled and observed for 12 months. Each participant undergoes a fluciclovine PET/CT scan as part of their normal clinical routine, with all images pseudonymized and stored in a central database where three independent nuclear medicine physicians, blinded to the local site's interpretation, review each scan. In addition to the initial imaging, follow-up assessments are conducted at one month and 12 months to validate scan findings; a questionnaire sent to the referring physician at one month helps capture any changes in the intended treatment plan, while comprehensive follow-up data-including additional imaging studies, PSA levels, treatment outcomes, and histopathological findings when available-are collected at 12 months. This follow-up information serves as a composite reference standard to distinguish true positive lesions from false positives, with criteria based on changes in lesion size, response to treatment, and confirmatory imaging or biopsy results, as well as to identify any false negatives.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male and aged >18 years old.
* Patient with a history of localized adenocarcinoma of the prostate with prior curative intent treatment, experiencing BCR of hormone sensitive PCa, following prior treatment with one or more of the following: a) RP, b) RP plus adjuvant therapy, c) RT and/or androgen deprivation therapy [ADT].
* An elevated PSA, clinically suspicious for biochemically recurrent disease, that meets one of the following conditions: 1) Following RP with or without adjuvant therapy: PSA ≥0.2 ng/mL followed by a subsequent confirmatory PSA value ≥0.2 ng/mL and within the total range of 0.2 and 2 ng/ml. PSA must be measured at least 6 weeks after RP. 2) Following RT (e.g. radical radiotherapy or brachytherapy) as the primary treatment: nadir +2 ng/mL and within the total range of 2 and 4 ng/ml

Exclusion Criteria:

* Patients with any medical condition or circumstance (including receiving an investigational product) that the investigator believes may compromise the data collected or lead to a failure to fulfill the study requirements.
* Current or recent androgen deprivation therapy (ADT) within 3 months prior to the start of the study, which includes surgical orchidectomy, continuous or intermittent LHRH agonist/antagonist, and first-/second-generation anti androgen alone or combined with LHRH agonist/antagonist.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a diagnosis of BCR and negative or inconclusive PSMA-ligand PET of previous radically treated PCa, aged ≥18 years old, eligible for fluciclovine PET/CT.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Patient-level detection rate | From enrollment to the end of observation at 1 year
  The patient-level detection rate of fluciclovine (18F) PET/CT in patients with a prior negative or inconclusive PSMA-ligand PET/CT

SECONDARY OUTCOMES:
Region level detection rate | From enrollment to the end of observation at 1 year
  Region level detection rate of fluciclovine (18F) PET/CT with prior negative or inconclusive PSMA-ligand PET/CT
Detection rate stratified by PSA level | From enrollment to the end of observation at 1 year
  Detection rate (patient and region level) of fluciclovine (18F) PET/CT with prior negative or inconclusive PSMA-ligand PET/CT, stratified by PSA level
Intended management change | From enrollment to the end of observation at 1 year
  The proportion of patients with a change of intended management after fluciclovine (18F) PET/CT
Interreader agreement | From enrollment to the end of observation at 1 year
  Reader kappa statistics of fluciclovine (18F) scan interpretation by the blinded independent readers

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Eiber, MD, Principal Investigator — Technical University of Munich
Locations (2):
- Germany (2):
  - University Hospital Augsburg, Augsburg, Bavaria
  - TUM University Hospital, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of anonymous data might be possible upon reasonable scientific request.